CLINICAL TRIAL: NCT03113643
Title: Phase 1 Study of SL-401 in Combination With Azacitidine and Venetoclax in Relapsed/Refractory Acute Myeloid Leukemia (AML) and in Treatment-Naive Subjects With AML Not Eligible for Standard Induction and in Subjects With Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN) or SL-401 in Combination With Azacitidine in Subjects With High-Risk Myelodysplastic Syndrome (MDS)
Brief Title: SL-401 in Combination With Azacitidine or Azacitidine/Venetoclax in Acute Myeloid Leukemia (AML), High-Risk Myelodysplastic Syndrome (MDS) or Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Stemline Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Andrew Lane, Andrew Lane, MD, PhD, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-056
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Blastic Plasmacytoid Dendritic Cell Neoplasm
Keywords: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Blastic Plasmacytoid Dendritic Cell Neoplasm; BPDCN
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Blastic Plasmacytoid Dendritic Cell Neoplasm | interventions — Azacitidine; tagraxofusp; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SL-401+ Azacitidine (Experimental): SL-401 will be administered every 4 weeks, on a 28 day cycle; SL-401 will be given intravenously; Azacitidine will be administered every 4 weeks, on a 28 day cycle; Azacitidine will be given intravenously or subcutaneously
  Interventions: Drug: Azacitidine; Drug: SL-401
- SL-401+ Azacitidine + Venetoclax (Experimental): SL-401 will be administered every 4 weeks, on a 28 day cycle; SL-401 will be given intravenously; Azacitidine will be administered every 4 weeks, on a 28 day cycle; Azacitidine will be given intravenously or subcutaneously; Venetoclax will be administered for 21 days on a 28 day cycle; Venetoclax will be taken orally
  Interventions: Drug: Azacitidine; Drug: SL-401; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Chemotherapy
  Other Names: Vidaza
Drug: SL-401 — SL-401 works by targeting leukemia cells (blasts), and also possibly by stopping or slowing the growth of cancer stem cells, which are the undeveloped cells which can develop into cancer cells.
Drug: Venetoclax — Venetoclax is a BH3-mimetic. Venetoclax blocks the anti-apoptotic B-cell lymphoma-2 (Bcl-2) protein, leading to programmed cell death of CLL cells. Overexpression of Bcl-2 in some lymphoid malignancies has sometimes shown to be linked with increased resistance to chemotherapy.
  Other Names: Venclyxto, Venclexta
  Arms: SL-401+ Azacitidine + Venetoclax

SUMMARY:
This research study is studying a drug as a possible treatment for diagnosis of AML, BPDCN and high-risk MDS.

The interventions involved in this study are:

* SL-401
* Azacitidine
* Venetoclax

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational intervention and also tries to define the appropriate dose of the investigational intervention to use for further studies. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has approved azacitidine and venetoclax as a treatment option for AML. However, the combination of these two drugs with SL-401 has not been FDA approved.

The combination of SL-401, azacitidine and venetoclax has not been FDA approved for BPDCN. However, SL-401 has been FDA approved for BPDCN.

The combination of SL-401 and azacitidine has not been FDA approved for BPDCN.

In this research study, the study drug SL-401 will be combined with the standard dose of azacitidine (for MDS patients) or azacitidine/venetoclax (for AML and BPDCN patients). The goal of this research study is to try and determine the safest, highest dose of study drug, SL-401, in combination with azacitidine or azacitidine/venetoclax that can be given to patients with AML, BPDCN or high-risk MDS. SL-401 works by stopping or slowing the growth of cancer stem cells, which are the undeveloped cells which can develop into cancer cells. The goals of this research study are to look at if this combination works to help treat your cancer and if there is any lasting effect of this combination. This study will also look at how the SL-401, in combination with azacitidine or azacitidine/venetoclax, affects certain proteins in your blood and bone marrow. SL-401 has been given to patients with AML, and MDS in the past, but this is the first time it will be given in combination with another drug.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed diagnosis of acute myeloid leukemia (AML) [Cohort B] or myelodysplastic syndrome (MDS) [Cohort A] or BPDCN [Cohort C] per 2016 WHO criteria

CD123 / IL3RA expression on the subject's AML or MDS blasts or BPDCN cells determined locally within 3 months of first protocol treatment

Age >= 18 years with relapsed or refractory AML (hydroxyurea is not considered a prior treatment regimen) [Cohort B]

OR

Age >= 18 years with treatment-naïve AML who decline intensive induction chemotherapy or who are unfit due to co-morbidity or other factors (see APPENDIX A for unfitness definitions) (hydroxyurea is not considered a prior treatment regimen) [Cohort B]

OR

Age >= 18 years with MDS and > 10% myeloblasts in the bone marrow [Cohort A]

OR

Age >= 18 years with relapsed or refractory BPDCN (hydroxyurea is not considered a prior treatment regimen) [Cohort C]

Adequate organ function as defined by:

Albumin > 3.2 g/dL (in the absence of receipt of intravenous albumin in the previous 72 hours) Serum creatinine < 1.5x ULN Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5x ULN Total bilirubin < 1.5x ULN (if thought to be > 1.5x ULN due to Gilbert's disease or the patient's AML, must discuss with the PI) Creatine phosphokinase (CPK) < 2.5x ULN Left ventricular ejection fraction > institutional lower limit of normal by MUGA scan or echocardiogram within 30 days of first protocol treatment

[Cohorts B and C] WBC < 20,000 / uL on day of first therapy, cytoreduction may be achieved using hydroxyurea

Ability to understand and the willingness to sign a written informed consent document.

Able to adhere to study visit schedule and other protocol requirements including follow-up for survival assessment

Women of child-bearing potential must agree to use adequate contraception for the duration of study participation and for 2 months after completion of protocol treatment.

Men treated or enrolled on this protocol must also agree to use adequate contraception for the duration of study participation and 2 months after completion of protocol treatment.

Exclusion Criteria:

Prior treatment with venetoclax [Cohorts B or C], unless it was last taken >2 months before protocol therapy

Diagnosis of acute promyelocytic leukemia

Received treatment with chemotherapy, radiation, or biologic cancer therapy within 14 days of first protocol treatment, except for intrathecal chemotherapy. Prior and concurrent hydroxyurea is permitted.

Hematopoietic stem cell transplantation (HSCT) within 60 days of screening or active graft versus-host-disease

Active CNS involvement by AML or BPDCN. Screening lumbar puncture (LP) required for patients with BPDCN. If history of treated CNS involvement, must have had two consecutive negative LPs since last CNS involvement, which may include the screening LP

Known positive status for HIV infection; known active hepatitis B or hepatitis C infection

Clinically significant cardiopulmonary disease including uncontrolled or NYHA class 3 or 4 congestive heart failure, uncontrolled angina, uncontrolled hypertension, uncontrolled arrhythmia, myocardial infarction or stroke within 6 months of first protocol treatment, or QTc > 480 ms

Patients with known active advanced malignant solid tumors are excluded (except for basal or squamous skin cancers, or carcinomas in situ). Patients with additional hematologic malignancies that require treatment are excluded.

Pregnant women are excluded from this study because there is an unknown but potential risk for adverse events in the developing fetus with SL-401, azacitidine, and venetoclax (negative urine or serum pregnancy test required within 14 days of Cycle 1, Day 1). Because nursing infants have unknown potential for adverse events secondary to treatment of the mother, breastfeeding should be discontinued if the mother is treated with SL-401, azacitidine, and venetoclax.

Patients with uncontrolled infection shall not be enrolled until infection is treated and brought under control. Patients with active infection are permitted to enroll provided that the infection is controlled

[Cohorts B and C] Patients with gastrointestinal (GI) tract disease causing the inability to take oral medication, malabsorption syndrome, a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's disease, ulcerative colitis)

[Cohorts B and C] Patients on strong CYP3A inducers within 7 days of first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2017-06-26 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 2 years
  To determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of SL-401 in combination with azacitidine or in combination with azacitidine and venetoclax in this patient population and evaluate the safety of this regimen

SECONDARY OUTCOMES:
Complete Response Rate | 2 years
  To estimate the complete remission (CR) / CR with incomplete count recovery (CRi) rate within 6 cycles of combination therapy consisting of SL-401 administered with azacitidine or in combination with azacitidine and venetoclax in subjects with AML and high-risk MDS
Time to response | 2 years
  To estimate the time to response with SL-401 in combination with azacitidine or in combination with azacitidine and venetoclax
Duration of remission | 2 years
  To estimate the duration of remission with SL-401 in combination with azacitidine or in combination with azacitidine and venetoclax
Progression Free Survival | 1 and 2 years
  To estimate the 1 and 2-year progression free survival (PFS) with SL-401 in combination with azacitidine or in combination with azacitidine and venetoclax
Overall Survival | 2 years
  To estimate the overall survival (OS) with SL-401 in combination with azacitidine or in combination with azacitidine and venetoclax

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Lane, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - City of Hope, Duarte, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lane AA, Garcia JS, Raulston EG, Garzon JL, Galinsky I, Baxter EW, Leonard R, DeAngelo DJ, Luskin MR, Reilly CR, Stahl M, Stone RM, Vedula RS, Wadleigh MM, Winer ES, Mughal T, Brooks C, Gupta IV, Stevenson KE, Neuberg DS, Ren S, Keating J, Konopleva M, Stein A, Pemmaraju N. Phase 1b trial of tagraxofusp in combination with azacitidine with or without venetoclax in acute myeloid leukemia. Blood Adv. 2024 Feb 13;8(3):591-602. doi: 10.1182/bloodadvances.2023011721. PMID 38052038
- [Derived] Wang SY, Thomassen K, Kurch L, Opitz S, Franke GN, Bach E, Platzbecker U, Kayser S. Combination of Tagraxofusp and Azacitidine Is an Effective Option for Relapsed Blastic Plasmacytoid Dendritic Cell Neoplasm After Allogeneic Hematopoietic Stem-Cell Transplantation. Clin Lymphoma Myeloma Leuk. 2021 Jul;21(7):e579-e582. doi: 10.1016/j.clml.2021.02.008. Epub 2021 Mar 2. No abstract available. PMID 33795208